CLINICAL TRIAL: NCT02887118
Title: Quantitative and Prognostic Evaluation of Dense Red Blood Cells in Sickle Cell Children: Single-center Study From the Creteil (France) Pediatric Cohort
Brief Title: Dense Red Blood Cells in Sickle Cell Children
Acronym: DREPADENSE
Status: Terminated | Type: Observational
Why Stopped: The recruiting centre was no longer presenting new patients for inclusion
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Corinne Pondarré, Doctor, Centre Hospitalier Intercommunal Creteil
Other Study IDs: DREPADENSE
Record Dates: First submitted 2016-06-21; First posted 2016-09-01 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Sickle Cell Disease
Keywords: Erythrocytes; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples to study dense red blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Common arm: Children with sickle cell anemia will be included. Blood samples of all the included patients will be collected during a day-hospitalization for a planned chek-up. For all these patients the number of dense erythrocytes will be evaluated

SUMMARY:
Quantitative and prognostic evaluation of dense red blood cells in sickle cell children: preliminary single center study from the Creteil pediatric cohort.

DETAILED DESCRIPTION:
An association between red blood cell density and hemolytic parameters, and clinical manifestations has been demonstrated in adults with sickle cell anemia.

This factor has not been studied in children. The identification of predictive biomarkers of disease severity, especially of specific pediatric complications (cerebral vasculopathy, splenic sequestration, Dactylitis) would be useful for optimal care of the children and early intensification Red blood cell density might be one of these prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 months-18 years
* Patient with sickle cell disease namely SS, or S / Beta0 or S / Beta +
* Patient regularly followed in the pediatric cohort of the CHI Creteil
* Patient Hospitalized for an annual check-up
* With or without intensification by Hydroxycarbamide
* patient who haven't been transfused within 3 months
* Whose parents have given their informed consent
* Patients insured to the French social scheme

Exclusion Criteria:

* Sickle cell SC disease
* Having received an allogeneic bone marrow transplantation
* Under regular transfusion program
* Having received a transfusion within 3 months

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with sickle cell disease followed regularly in the CHI creteil hospital aged from 18 months to 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
number of dense red blood cells (DRBC) | 1 day
  Evaluation of the number of dense red blood cells in the blood of affected children

SECONDARY OUTCOMES:
biological profile | 1 day
  hemolytic parameters (LDH, bilirubin, Hemoglobin level)
Number of patients with velocities > 200 cm/sec on transcranial doppler | 1 day
  Cerebral vasculopathy (correlation with patients with abnormal velocities on transcranial doppler (TCD)(> 200 cm/sec)
  History of dactylitis History of ischemic lesions on magnetic resonance imaging (MRI)
Number of patients with history of acute splenic sequestration, | 1 day
Number of patients with history of acute chest syndrome | 1 day
Number of patients with History of dactylitis | 1 day
Number of patients with history of abnormal transcranial doppler (TCD) (≥ 200 cm/sec) | 1 day
Number of patients with history of ischemic lesions on magnetic resonance imaging (MRI) | 1 day
Number of patients with hydroxycarbamide treatment | 1 day
  effect of hydroxycarbamide on the % DRBC
Number of dense red blood cells | 1 day
  number of dense red blood cells in the pediatric population with no known blood condition

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Pondarre, MD PhD, Principal Investigator — CHI Créteil
Locations (1):
- CHI Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller ST, Sleeper LA, Pegelow CH, Enos LE, Wang WC, Weiner SJ, Wethers DL, Smith J, Kinney TR. Prediction of adverse outcomes in children with sickle cell disease. N Engl J Med. 2000 Jan 13;342(2):83-9. doi: 10.1056/NEJM200001133420203. PMID 10631276
- [Background] Benkerrou M, Alberti C, Couque N, Haouari Z, Ba A, Missud F, Boizeau P, Holvoet L, Ithier G, Elion J, Baruchel A, Ducrocq R. Impact of glucose-6-phosphate dehydrogenase deficiency on sickle cell anaemia expression in infancy and early childhood: a prospective study. Br J Haematol. 2013 Dec;163(5):646-54. doi: 10.1111/bjh.12590. Epub 2013 Oct 10. PMID 24117340
- [Background] Quinn CT, Shull EP, Ahmad N, Lee NJ, Rogers ZR, Buchanan GR. Prognostic significance of early vaso-occlusive complications in children with sickle cell anemia. Blood. 2007 Jan 1;109(1):40-5. doi: 10.1182/blood-2006-02-005082. Epub 2006 Aug 29. PMID 16940426
- [Background] Bernaudin F, Verlhac S, Arnaud C, Kamdem A, Chevret S, Hau I, Coic L, Leveille E, Lemarchand E, Lesprit E, Abadie I, Medejel N, Madhi F, Lemerle S, Biscardi S, Bardakdjian J, Galacteros F, Torres M, Kuentz M, Ferry C, Socie G, Reinert P, Delacourt C. Impact of early transcranial Doppler screening and intensive therapy on cerebral vasculopathy outcome in a newborn sickle cell anemia cohort. Blood. 2011 Jan 27;117(4):1130-40; quiz 1436. doi: 10.1182/blood-2010-06-293514. Epub 2010 Nov 10. PMID 21068435
- [Background] Bartolucci P, Brugnara C, Teixeira-Pinto A, Pissard S, Moradkhani K, Jouault H, Galacteros F. Erythrocyte density in sickle cell syndromes is associated with specific clinical manifestations and hemolysis. Blood. 2012 Oct 11;120(15):3136-41. doi: 10.1182/blood-2012-04-424184. Epub 2012 Aug 23. PMID 22919030
- [Background] Thornburg CD, Files BA, Luo Z, Miller ST, Kalpatthi R, Iyer R, Seaman P, Lebensburger J, Alvarez O, Thompson B, Ware RE, Wang WC; BABY HUG Investigators. Impact of hydroxyurea on clinical events in the BABY HUG trial. Blood. 2012 Nov 22;120(22):4304-10; quiz 4448. doi: 10.1182/blood-2012-03-419879. Epub 2012 Aug 22. PMID 22915643
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083